CLINICAL TRIAL: NCT05938335
Title: Results of Sequencing of a Large Panel of Genes From Leptin Melanocortin Pathway in Children Suffering From Severe Obesity
Brief Title: Sequencing of 14 Genes From Leptin Melanocortin Pathway in Severe Obesity in Childhood.
Acronym: OBEGEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENARD Emeline, Doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023PI
Record Dates: First submitted 2023-06-12; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Obesity, Child
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- severe obese children (Experimental): children with severe obesity with BMI > 3sds
  Interventions: Genetic: sequencing of a panel of 14 genes in leptin melanocortin pathway

INTERVENTIONS:
Genetic: sequencing of a panel of 14 genes in leptin melanocortin pathway — sequencing (NGS) of a panel of 14 genes in leptin melanocortin pathway in french children with severe obesity

SUMMARY:
About 380 million children and adolescents suffer from overweight and obesity at the global level. Obesity results from the interplay between biological (sex, age, fetal programming, gut microbiota, epigenetics, and genetics) and environmental factors (e.g., unhealthy diet, physical inactivity, stress). Mutations in genes from leptin melanocortin pathway are involved in "non syndromic monogenic obesity", characterized by severe early onset obesity, hyperphagia and endocrine deficiencies. Exact frequencies of mutation in these genes are not precisely evaluated in french children with severe obesity. Moreover new treatment, such seltmelanotide are avalaible in case of certain mutation, leading to a significative weight loss in treated patients.

DETAILED DESCRIPTION:
Obesity is a global health concern that affected more than 650 million adult people and more than 380 million children and adolescents worldwide, with no signs of slowing down despite major investments in health policy. Obestiy is a multifactorial disease, but 40 to 75% of body mass index (BMI) variation is explained by genetic factors.

Mutations in genes from leptin melanocortin pathway lead to "non syndromic monogenic obesity", characterized by severe early onset obesity, hyperphagia and endocrine deficiencies. This pathway plays a central role in regulating mammalian food intake, energy expenditure and body weight regulation. Somes genes are well characterized such LEP gene, LEPR gene, or MC4R but others have been recently described as ADCY3, SIM1, SH2B1, NTRK2, BDNF, KSR2.

The frequency of these mutations are not precisely estimated in a group of french children with severe obesity.

Moreover, a precocious identification of these mutations, could afford, in certain case the possibility of a efficient treatment with setmelanotide, leading to a significant weight loss in treated patients.

ELIGIBILITY:
Inclusion Criteria:

* severe obesity with BMI > 3SDS

Exclusion Criteria:

* genetic obesity (Prader Willi syndrome, Bardet Biedl syndrome, X fragile syndrome, Alstrom syndrome)
* BMI < 3 SDS
* age < 6 months
* monogenic non syndromic obesity, with mutation in genes of leptin melanocortin pathway previously diagnosed
* cushing syndrome

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
frequency of mutations of genes from leptin melanocortin pathway | 1 year
  Evaluating of the frequency of mutations of 14 genes from leptin melanocortin pathway (LEP, LEPR, POMC, PCSK1, MC3R, MC4R, MRAP2, ADCY3, SIM1, SH2B1, NTRK2, BDNF, KSR2) in a group of french children with severe obesity.

SECONDARY OUTCOMES:
Clinical characteristics of children with severe obesity followed in CHRU of Nancy | 1 year
  Description of the clinical characteristics : height in cm BMI
Clinical characteristics of children with mutations of leptin melanocortin pathway | 1 year
  Description of the clinical characteristics :thyroid function (TSH T3 T4)
Clinical characteristics of children with mutations of leptin melanocortin pathway | 1 year
  Description of the clinical characteristics : IGF1 levels
Clinical characteristics of children with mutations of leptin melanocortin pathway | 1 year
  Description of the clinical characteristics :BMI in kg/m²
Clinical characteristics of children with mutations of leptin melanocortin pathway | 1 year
  Description of the clinical characteristics : weight in kg
Clinical characteristics of children with mutations of leptin melanocortin pathway | 1 year
  Description of the clinical characteristics : bone age (X ray of the left hand)
Clinical characteristics of children with mutations of leptin melanocortin pathway | 1 year
  Description of the clinical characteristics : metabolic profile
Clinical characteristics of children with mutations of leptin melanocortin pathway | 1 year
  Description of the clinical characteristics : leptin level
Penetrance of mutations from leptin melanocortin pathway | 1 year
  Evaluation of the penetrance of mutation from leptin melanocortin pathway, that is to say the percentage of obesity in mutation carrier
effect of age, sex, country of birth on mutations' penetrance. | 1 year
  Evaluation of the effect of age, sex, country of birth on mutations' penetrance.
Clinical characteristics of children with severe obesity followed in CHRU of Nancy | 1 year
  Description of Clinical characteristics of children with severe obesity followed in CHRU of Nancy : weight in kg Description of the clinical characteristics :
Clinical characteristics of children with severe obesity followed in CHRU of Nancy | 1 year
  Description of the clinical characteristics :BMI in kg/m²

IPD SHARING:
Plan to Share IPD: Undecided